CLINICAL TRIAL: NCT06910683
Title: Technology dRiven Enhancement to Engage & Connect
Acronym: TREE-Connect
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-04027370
Record Dates: First submitted 2025-03-18; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREE-Connect + Clinician-delivered psychotherapy (Experimental): Participants will receive a hybrid intervention that includes clinician-delivered psychotherapy and a TREE-Connect app
  Interventions: Behavioral: TREE-Connect; Behavioral: Clinician-delivered psychotherapy
- Clinician-delivered psychotherapy (Active Comparator): Participants will receive clinician-delivered psychotherapy without the TREE-Connect app
  Interventions: Behavioral: Clinician-delivered psychotherapy

INTERVENTIONS:
Behavioral: TREE-Connect — TREE-Connect is a mental health app that aims to increase engagement in rewarding activities
  Arms: TREE-Connect + Clinician-delivered psychotherapy
Behavioral: Clinician-delivered psychotherapy — Clinician-delivered psychotherapy is delivered remotely and aimed to increase engagement in rewarding activities

SUMMARY:
This study will investigate whether an intervention that includes remotely delivered therapy sessions and a digital mental health app, compared to only remotely delivered therapy reduces late-life depression

DETAILED DESCRIPTION:
Depression in mid- and late-life is characterized with reduced functions of the reward system. The investigators designed a psychotherapy that aims to improve reward functions through engagement in pleasurable activities and in turn reduce depression. Prior work has shown that this therapy is acceptable and reduces depression. This study examines whether a hybrid intervention that combines clinician remotely-delivered psychotherapy, and a novel app named TREE-Connect, reduces late life depression. This TREE-Connect app uses a machine learning algorithm to promote adherence to therapy (completion of therapeutic homework) in late-life depression and increase cost-effectiveness and reach of treatment to older adults. This randomized controlled trials will test whether the hybrid intervention (clinician-delivered psychotherapy + app), compared to a condition that includes solely clinician-delivered therapy is acceptable and reduces late-life depression.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50-80
* Capacity to provide consent for research assessment and treatment.
* Significant depression, i.e., PHQ-9 ≥10 (moderate severity of symptoms)
* Mini Mental Status Exam (MMSE) equal or greater than a score of 23.
* Off antidepressants or on stable dose for 8 weeks and do not intend to change the dose in the next 10 weeks, without individual psychotherapy services during the study period.

Exclusion Criteria:

* Intent or plan to commit suicide in the near future.
* Inability to communicate in English.
* History or presence of psychiatric diagnoses other than major depressive disorder without psychotic features, generalized anxiety disorder, specific phobia, or antisocial or borderline personality disorder.
* Neurological disorders (dementias, amnestic and multidomain Mild Cognitive Impairment, Parkinson's disease, epilepsy, etc.).
* Acute or severe medical illness in the past 3 months (metastatic cancer, multiple sclerosis, decompensated cardiac, liver or kidney failure, major surgery, stroke or myocardial infarction, cardiac, renal, or respiratory failure; severe chronic obstructive pulmonary disease, etc.) that may be the primary cause depressive symptoms, influence brain systems of interest, or impact ability to participate in the study.
* For MRI only: Contraindications to MRI scanning including cardiac pacemaker, heart valve replacement, vascular stent, insulin pump, cochlear implant, any other metallic biomedical implant contraindicating to MRI, and claustrophobia.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability (Client Satisfaction Questionnaire; CSQ) | 9 Weeks
  Acceptability will measured using the Client Satisfaction Questionnaire (CSQ) with a benchmar score of >=3 (out of 4; average score); Range: 0 to 4, with higher scores indicating greater acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Nili Solomonov, PhD, Principal Investigator — Weill Medical College of Cornell University; Samprit Banerjee, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Relevant de-identified data as well as study protocol, treatment manuals, statistical analysis plan and informed consent.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Available to researchers upon reasonable request
Access Criteria: Available to researchers upon reasonable request